CLINICAL TRIAL: NCT06653803
Title: Ultrasound-guided Rhomboid Intercostal Block Versus Retrolaminar Block for Postoperative Analgesia After Thoracoscopic Sympathectomy: A Randomized Clinical Trial
Brief Title: Rhomboid Intercostal Block Versus Retrolaminar Block for Postoperative Analgesia After Thoracoscopic Sympathectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour Teaching Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DTH: 24001
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-07

CONDITIONS: Post Operative Pain
Keywords: Rhomboid Intercostal Block; Retrolaminar Block; Regional Analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (n=30) (Active Comparator): Rhomboid Intercostal Block
  Interventions: Procedure: Rhomboid Intercostal Block (RIB)
- Group B (n=30) (Active Comparator): Retrolaminar Block
  Interventions: Procedure: Retrolaminar Block (RLB)

INTERVENTIONS:
Procedure: Rhomboid Intercostal Block (RIB) — Intraoperative Ipsilateral Ultrasound-guided RIB
  Arms: Group A (n=30)
Procedure: Retrolaminar Block (RLB) — Intraoperative Ipsilateral Ultrasound-guided RLB
  Arms: Group B (n=30)

SUMMARY:
Background: Although thoracoscopic sympathectomy is made via small incisions, it is associated with severe postoperative pain. Both Rhomboid intercostal block (RIB) and Retrolaminar block (RLB) are recent techniques used for pain control after such procedures

Objectives: To compare the effectiveness of RIB and RLB in providing postoperative analgesia after thoracoscopic sympathectomy in adult patients and their impact on the patient's outcomes.

Patients and Methods: This prospective, randomized (1:1), double-blind clinical trial; will be carried out on 60 patients scheduled for elective thoracoscopic sympathectomy under general anesthesia at our hospital. Patients will be randomly allocated into two equal groups (30 patients each) and will receive: in group A; general anesthesia with intraoperative ipsilateral ultrasound-guided RIB, whereas in group B; general anesthesia with intraoperative ipsilateral ultrasound-guided RLB.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status ≤ II
* Age from 18 to 60 years
* Body Mass Index (BMI) < 35 kg/m²

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status > II
* Age < 18 years or > 60 years
* Body Mass Index (BMI) ≥ 35
* Local infection at the puncture site
* Altered mental status
* Pregnant women
* Allergy to study drugs
* Chronic pain
* Coagulation abnormalities or on anticoagulants
* Severe hepatic or kidney disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Mean and Standard deviation of time to the first request of postoperative rescue analgesic (minutes) (mean±SD) | 24 hours after the end of surgery
  The time interval between the block performance and the first request of postoperative analgesia

SECONDARY OUTCOMES:
Mean and Standard deviation of Numeric Pain Rating Scale (NPRS) score (mean±SD) | 24 hours after the end of surgery
  NPRS measures the severity of postoperative pain, it is a 11 point scale from 0-10; where 0=No pain and 10=Worst possible pain (At PACU, 1h, 3h, 6h, 12h, 18h, 24h) after the end of surgery
Mean and Standard deviation of the total dose of the rescue analgesic consumed (milligrams) (mean±SD) | 24 hours after the end of surgery
  The total dose of the rescue analgesic consumed in the first 24 hours after the end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Shaat, MD, Principal Investigator — Damanhour Teaching Hospital
Locations (1):
- Damanhour Teaching Hospital, Damanhūr, El-Beheira, Egypt